CLINICAL TRIAL: NCT01737398
Title: A Phase 2/3 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of ISIS 420915 in Patients With Familial Amyloid Polyneuropathy (NEURO-TTR Study)
Brief Title: Efficacy and Safety of Inotersen in Familial Amyloid Polyneuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 420915-CS2
Expanded Access: NCT03400098 (Approved for marketing)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
Keywords: FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis | interventions — Inotersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inotersen (Active Comparator): 300 mg inotersen administered subcutaneously (SC) 3 times on alternate days in the first week and then once-weekly for 64 weeks
  Interventions: Drug: Inotersen
- Placebo (Active Comparator): Placebo administered SC 3 times on alternate days in the first week and then once-weekly for 64 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inotersen
  Other Names: TEGSEDI; IONIS-TTR Rx; ISIS 420915
  Arms: Inotersen
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of inotersen given for 65 weeks in participants with Familial Amyloid Polyneuropathy (FAP).

DETAILED DESCRIPTION:
FAP is a rare, hereditary disease caused by mutations in the transthyretin (TTR) protein. TTR is made by the liver and secreted into the blood. TTR mutations cause it to misfold and deposit in multiple organs causing FAP.

Inotersen (also known as ISIS 420915) is an antisense drug that was designed to decrease the amount of mutant and normal TTR made by the liver. It is predicted that decreasing the amount of TTR protein would result in a decrease in the formation of TTR deposits, and thus slow or stop disease progression.

The purpose of this study is to determine if inotersen can slow or stop the nerve damage caused by TTR deposits. This study will enroll late Stage 1 and early Stage 2 FAP participants. Participants will receive either inotersen or placebo for 65 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 and Stage 2 FAP participants with the following:

  1. NIS score within protocol criteria
  2. Documented transthyretin variant by genotyping
  3. Documented amyloid deposit by biopsy
* Females of child-bearing potential must use appropriate contraception and be non-pregnant and non-lactating. Males engaging in relations of child-bearing potential are to use appropriate contraception

Exclusion Criteria:

* Low Retinol level at screen
* Karnofsky performance status ≤50
* Poor Renal function
* Known type 1 or type 2 diabetes mellitus
* Other causes of sensorimotor or autonomic neuropathy (for example, autoimmune disease)
* If previously treated with Vyndaqel®, will need to have discontinued treatment for 2 weeks prior to Study Day 1. If previously treated with Diflunisal, will need to have discontinued treatment for 3 days prior to Study Day 1
* Previous treatment with any oligonucleotide or siRNA within 12 months of screening
* Prior liver transplant or anticipated liver transplant within 1 year of screening
* New York Heart Association (NYHA) functional classification of ≥3
* Acute Coronary Syndrome or major surgery within 3 months of screening
* Known Primary or Leptomeningeal Amyloidosis
* Anticipated survival less than 2 years
* Any other conditions in the opinion of the investigator which interfere with the participant participating in or completing the study

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (9):
  - University of California, Irvine, Orange, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University Bayview Medical Center, Baltimore, Maryland
  - Boston University School of Medicine - Amyloid Treatment & Research Program, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center - The Neurological Institute, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
- FLENI, Buenos Aires, Argentina
- Brazil (3):
  - Federal University of Rio de Janeiro - University Hospital, Rio de Janeiro
  - AACD, São Paulo
  - UNIFESP, São Paulo
- France (2):
  - CHU Henri Mondor - Department of Neurology, Créteil
  - CHU Bicetre Aphp French Referral Center for FAP/Cornamyl Network, Le Kremlin-Bicêtre
- UKM; Universitätsklinikum Münster, Klinik für Transplantationsmedizin, Münster, Germany
- Italy (2):
  - Universita Degli Studi Di Messina - Azienda Ospedaliera Universitaria Policlinico "Gaetano Martino", Messina, Sicily
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico San Matteo, Pavia
- Auckland City Hospital, Auckland, New Zealand
- Portugal (2):
  - CHLN - Hospital de Santa Maria, Lisbon
  - CHP-HGSA, Unidade Clinica de Paramiloidose, Porto
- Spain (2):
  - Hospital Universitari Vall D' Hebron, Barcelona
  - Hospital Clínic, Barcelona
- University College London - National Amyloidosis Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benson MD, Waddington-Cruz M, Berk JL, Polydefkis M, Dyck PJ, Wang AK, Plante-Bordeneuve V, Barroso FA, Merlini G, Obici L, Scheinberg M, Brannagan TH 3rd, Litchy WJ, Whelan C, Drachman BM, Adams D, Heitner SB, Conceicao I, Schmidt HH, Vita G, Campistol JM, Gamez J, Gorevic PD, Gane E, Shah AM, Solomon SD, Monia BP, Hughes SG, Kwoh TJ, McEvoy BW, Jung SW, Baker BF, Ackermann EJ, Gertz MA, Coelho T. Inotersen Treatment for Patients with Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):22-31. doi: 10.1056/NEJMoa1716793. PMID 29972757
- [Derived] Karam C, Brown D, Yang M, Done N, Zhu JJ, Greatsinger A, Bozas A, Vera-Llonch M, Signorovitch J. Long-term treatment effects of inotersen on health-related quality of life in patients with hATTR amyloidosis with polyneuropathy: Analysis of the open-label extension of the NEURO-TTR trial. Muscle Nerve. 2022 Oct;66(4):438-446. doi: 10.1002/mus.27675. Epub 2022 Aug 4. PMID 35799473
- [Derived] Karam C, Brown D, Yang M, Done N, Dieye I, Bozas A, Vera Llonch M, Signorovitch J. Factors associated with increased health-related quality-of-life benefits in hereditary transthyretin amyloidosis polyneuropathy patients treated with inotersen. Muscle Nerve. 2022 Sep;66(3):319-328. doi: 10.1002/mus.27668. Epub 2022 Jul 15. PMID 35766224
- [Derived] Yarlas A, Lovley A, McCausland K, Brown D, Vera-Llonch M, Conceicao I, Karam C, Khella S, Obici L, Waddington-Cruz M. Early Data on Long-term Impact of Inotersen on Quality-of-Life in Patients with Hereditary Transthyretin Amyloidosis Polyneuropathy: Open-Label Extension of NEURO-TTR. Neurol Ther. 2021 Dec;10(2):865-886. doi: 10.1007/s40120-021-00268-x. Epub 2021 Aug 5. PMID 34355354
- [Derived] Yarlas A, Lovley A, Brown D, Kosinski M, Vera-Llonch M. Responder analysis for neuropathic impairment and quality-of-life assessment in patients with hereditary transthyretin amyloidosis with polyneuropathy in the NEURO-TTR study. J Neurol. 2022 Jan;269(1):323-335. doi: 10.1007/s00415-021-10635-1. Epub 2021 Jun 14. PMID 34125267
- [Derived] Yu RZ, Wang Y, Norris DA, Kim TW, Narayanan P, Geary RS, Monia BP, Henry SP. Immunogenicity Assessment of Inotersen, a 2'-O-(2-Methoxyethyl) Antisense Oligonucleotide in Animals and Humans: Effect on Pharmacokinetics, Pharmacodynamics, and Safety. Nucleic Acid Ther. 2020 Oct;30(5):265-275. doi: 10.1089/nat.2020.0867. Epub 2020 Aug 19. PMID 32833564
- [Derived] Dyck PJB, Kincaid JC, Wiesman JF, Polydefkis M, Litchy WJ, Mauermann ML, Ackermann EJ, Guthrie S, Pollock M, Jung SW, Baker BF, Dyck PJ. mNIS+7 and lower limb function in inotersen treatment of hereditary transthyretin-mediated amyloidosis. Muscle Nerve. 2020 Oct;62(4):502-508. doi: 10.1002/mus.27022. Epub 2020 Aug 13. PMID 32654212
- [Derived] Dyck PJB, Coelho T, Waddington Cruz M, Brannagan TH 3rd, Khella S, Karam C, Berk JL, Polydefkis MJ, Kincaid JC, Wiesman JF, Litchy WJ, Mauermann ML, Ackermann EJ, Baker BF, Jung SW, Guthrie S, Pollock M, Dyck PJ. Neuropathy symptom and change: Inotersen treatment of hereditary transthyretin amyloidosis. Muscle Nerve. 2020 Oct;62(4):509-515. doi: 10.1002/mus.27023. Epub 2020 Aug 7. PMID 32654156
- [Derived] Coelho T, Yarlas A, Waddington-Cruz M, White MK, Sikora Kessler A, Lovley A, Pollock M, Guthrie S, Ackermann EJ, Hughes SG, Karam C, Khella S, Gertz M, Merlini G, Obici L, Schmidt HH, Polydefkis M, Dyck PJB, Brannagan Iii TH, Conceicao I, Benson MD, Berk JL. Inotersen preserves or improves quality of life in hereditary transthyretin amyloidosis. J Neurol. 2020 Apr;267(4):1070-1079. doi: 10.1007/s00415-019-09671-9. Epub 2019 Dec 18. PMID 31853709
- [Derived] Pinto MV, Dyck PJB, Gove LE, McCauley BM, Ackermann EJ, Hughes SG, Waddington-Cruz M, Dyck PJ. Kind and distribution of cutaneous sensation loss in hereditary transthyretin amyloidosis with polyneuropathy. J Neurol Sci. 2018 Nov 15;394:78-83. doi: 10.1016/j.jns.2018.08.031. Epub 2018 Aug 30. PMID 30219500
- [Derived] Waddington-Cruz M, Ackermann EJ, Polydefkis M, Heitner SB, Dyck PJ, Barroso FA, Wang AK, Berk JL, Dyck PJB, Monia BP, Hughes SG, Tai L, Jesse Kwoh T, Jung SW, Coelho T, Benson MD, Gertz MA. Hereditary transthyretin amyloidosis: baseline characteristics of patients in the NEURO-TTR trial. Amyloid. 2018 Sep;25(3):180-188. doi: 10.1080/13506129.2018.1503593. Epub 2018 Aug 31. PMID 30169969

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized: 113 inotersen and 60 placebo; received study treatment: 112 inotersen and 60 placebo. This study consisted of a 65-week Treatment Period, 1-week End of Treatment (EOT) Period, and a 6-month Post-treatment Evaluation Period.
Groups:
- Inotersen: Participants received 3 subcutaneous (SC) doses of 300 milligrams (mg) inotersen during Week 1, followed by once-weekly SC administration for 64 weeks.
- Placebo: Participants received 3 SC doses of placebo during Week 1, followed by once-weekly SC administration for 64 weeks.
Period: Overall Study
Arm/Group | Inotersen | Placebo
Started | 113 | 60
Received at Least 1 Dose of Study Drug (One participant in the inotersen group was ineligible, but was randomized in error.) | 112 | 60
Safety Set | 112 | 60
Completed | 87 | 52
Not Completed | 26 | 8
Not completed — Adverse event or SAE | 16 | 1
Not completed — Stopping rule met | 2 | 1
Not completed — Voluntary withdrawal | 2 | 3
Not completed — Ineligibility | 1 | 0
Not completed — Liver transplant | 1 | 0
Not completed — Disease progression | 2 | 3
Not completed — Sponsor's decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: Participants who were randomized and received at least 1 dose of study drug (inotersen or placebo). The Safety Set is the population used for the analyses of all safety measures.
Groups:
- Inotersen: Participants received 3 SC doses of 300 mg inotersen during Week 1, followed by once-weekly SC administration for 64 weeks.
- Total: Total of all reporting groups
Arm/Group | Inotersen | Placebo | Total
Number analyzed (Participants) | 112 | 60 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.53) | 59.5 (14.05) | 59.2 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 19 | 54
  Male | 77 | 41 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 7 | 24
  Not Hispanic or Latino | 95 | 53 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  Black | 3 | 1 | 4
  White | 105 | 53 | 158
  White & Grayish-Brown | 0 | 1 | 1
  Other | 3 | 2 | 5
Participants diagnosed with hATTR-CM [Count of Participants; unit: Participants]
  Yes | 45 | 22 | 67
  No | 67 | 38 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In The Modified Neuropathy Impairment Score (mNIS) +7 Composite Score at Week 66
Description: The mNIS+7 composite score is a measure of neurologic impairment that evaluates muscle weakness, sensation, reflexes, nerve conduction, and autonomic function. The mNIS+7 Composite Score has a range of -22.32 to 346.32 and a higher mNIS+7 composite score indicates lower function.
Time Frame: Baseline and Week 66
Population: The full analysis set included all randomized participants who received at least 1 injection of study drug (inotersen or placebo) and who had a Baseline and at least 1 post-Baseline efficacy assessment for the mNIS+7 score or Norfolk QoL-DN questionnaire total score. Participants analyzed = participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 85 | 52
Scores on a Scale | 4.16 (15.672) | 23.89 (24.190)
Statistical Analysis 1: Comparison: Inotersen vs Placebo; Test type: Other; p = 0.00000004, MMRM; Least Square Mean Difference = -19.73, 95% CI 2-sided [-26.43 to -13.03]

2. Primary Outcome: Change From Baseline In The Norfolk Quality Of Life Diabetic Neuropathy (QoL-DN) Questionnaire at Week 66
Description: The Norfolk QoL-DN score is a measure of physical function/large fiber neuropathy, symptoms, activities of daily living, small fiber neuropathy, and autonomic neuropathy. The Norfolk QoL-DN total score has a range of -4 to 136, and a higher Norfolk QoL-DN score indicates poorer QoL.
Time Frame: Baseline and Week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 84 | 52
Scores on a Scale | -0.08 (18.967) | 10.77 (21.134)
Statistical Analysis 1: Comparison: Inotersen vs Placebo; Test type: Other; p = 0.0006, MMRM; Least Square Mean Difference = -11.68, 95% CI 2-sided [-18.29 to -5.06]

3. Secondary Outcome: Change From Baseline In The Norfolk QoL-DN Questionnaire Symptoms Domain Score at Week 66
Description: The Norfolk QoL-DN symptoms score is a sub-score of the total Norfolk QoL-DN Questionnaire. The Norfolk QoL-DN symptoms domain score has a range of 0-32, and a higher Norfolk QoL-DN score indicates poorer QoL.
Time Frame: Baseline and Week 66
Population: This endpoint only measured participants with Stage 1 hATTR-PN in Full Analysis Set. Participants analyzed = participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 55 | 33
Scores on a Scale | -1.40 (4.763) | 1.18 (5.270)

4. Secondary Outcome: Change From Baseline In The Norfolk QoL-DN Questionnaire Physical Functioning/Large Fiber Neuropathy Domain Score at Week 66
Description: The Norfolk QoL-DN physical functioning/large fiber neuropathy domain score is a sub-score of the total Norfolk QoL-DN Questionnaire. The Norfolk QoL-DN physical function/large fiber neuropathy domain score has a range of -4 to 56, and a higher Norfolk QoL-DN domain score indicates poorer QoL.
Time Frame: Baseline and Week 66
Population: This endpoints only measured participants who had Stage 2 hATTR-PN in Full Analysis Set. Participants analyzed = participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 29 | 19
Scores on a Scale | 1.05 (11.924) | 8.74 (9.689)

5. Secondary Outcome: Change From Baseline In Modified Body Mass Index (mBMI) at Week 65
Description: The mBMI is the BMI multiplied by the serum albumin g/L
Time Frame: Baseline and Week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2*g/L
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 82 | 49
kg/m^2*g/L | -73.32 (96.311) | -85.21 (91.259)

6. Secondary Outcome: Change From Baseline In Body Mass Index (BMI) at Week 65
Time Frame: Baseline and Week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 82 | 49
kg/m^2 | -0.24 (1.521) | -0.87 (1.202)

7. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 66
Description: The NIS score is a measure of neurologic impairment. The NIS Score has a range of 0 to 244 and a higher NIS score indicates lower function.
Time Frame: Baseline and Week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 85 | 52
Scores on a Scale | 4.47 (10.329) | 17.29 (16.986)

8. Secondary Outcome: Change From Baseline in Modified +7 at Week 66
Description: The Modified +7 score is a version of the NIS score that is a measure of neurologic impairment. The Modified +7 Score has a range of -22.32 to 102.32 and a higher NIS score indicates lower function.
Time Frame: Baseline and Week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 85 | 52
Scores on a Scale | -0.31 (11.134) | 6.60 (12.770)

9. Secondary Outcome: Change From Baseline in NIS+7 at Week 66
Description: The NIS+7 score is a version of the NIS score that is a measure of neurologic impairment. The NIS+7 Score has a range of -26.04 to 270.04 and a higher NIS score indicates lower function.
Time Frame: Baseline and Week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 85 | 52
Scores on a Scale | 5.10 (10.709) | 19.00 (16.824)

10. Secondary Outcome: Change From Baseline in Global Longitudinal Strain (GLS) by Echocardiogram (ECHO) at Week 65 in the CM-ECHO Set
Description: GLS by ECHO is a measure of cardiac systolic function
Time Frame: Baseline and Week 65
Population: The CM-ECHO Set includes the subset of the Randomized Set who had a diagnosis of TTR cardiomyopathy at study entry but are not in the ECHO subgroup, plus participants who qualified to participate in the ECHO subgroup (whether consented or not). Participants analyzed = participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 50 | 25
Percent Change | 0.69 (3.134) | 0.46 (2.702)

11. Secondary Outcome: Change From Baseline in Global Longitudinal Strain (GLS) by Echocardiogram ECHO at Week 65 in the ECHO Subgroup
Description: GLS by ECHO is a measure of cardiac systolic function
Time Frame: Baseline and Week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 30 | 16
Percent Change | 0.25 (3.163) | 1.05 (2.745)

12. Secondary Outcome: Change From Baseline in Transthyretin (TTR) Level at Week 65
Time Frame: Baseline and Week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 84 | 51
g/L | -0.1570 (0.0619) | -0.0146 (0.0402)

13. Secondary Outcome: Change From Baseline in Retinol Binding Protein 4 (RBP4) Level at Week 65
Time Frame: Baseline and Week 65
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Inotersen | Placebo
Number analyzed (Participants) | 83 | 51
ug/L | -21725.9 (9884.04) | -1768.7 (8027.78)

14. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) Of Inotersen At Week 65
Time Frame: Week 65
Population: The PK Set was defined as all randomized participants who received at least 1 dose of active study drug (inotersen) and had at least 1 evaluable PK sample collected and analyzed with a reportable result.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Inotersen 300 mg IM Negative: Participants received 3 SC doses of 300 mg inotersen during Week 1, followed by once-weekly SC administration for 64 weeks, and had a negative immunogenicity (IM) status.
- Inotersen 300 mg IM Positive: Participants received 3 SC doses of 300 mg inotersen during Week 1, followed by once-weekly SC administration for 64 weeks, and had a positive IM status.
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 5 | 3
ug/mL | 6.76 (1.88) | 11.1 (4.80)

15. Secondary Outcome: Time To The Maximum Plasma Concentration (Tmax) Of Inotersen At Week 65
Time Frame: Week 65
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Inotersen 300 mg IM Negative: Participants received 3 SC doses of 300 mg inotersen during Week 1, followed by once-weekly SC administration for 64 weeks, and had a negative IM status.
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 5 | 3
hours | 4.14 (1.88) | 3.48 (0.68)

16. Secondary Outcome: Area Under The Plasma Concentration-time Curve From 0 To 24 Hours (AUC[0-24hr]) Of Inotersen At Week 65
Time Frame: Week 65
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 5 | 3
ug*hr/mL | 93.1 (30.7) | 92.4 (77.3)

17. Secondary Outcome: Area Under The Plasma Concentration-time Curve From 0 To 168 Hours (AUC[0-168hr]) Of Inotersen At Week 65
Time Frame: Week 65
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 4 | 3
ug*hr/mL | 98.9 (33.5) | 103.0 (88.2)

18. Secondary Outcome: Plasma Clearance From 0 To 24 Hours (CL[0-24hr]/F) Of Inotersen At Week 65
Time Frame: Week 65
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 5 | 3
L/hr | 3.57 (1.32) | 6.14 (5.92)

19. Secondary Outcome: Inotersen Plasma Clearance At Steady State (CLss/F) At Week 65
Time Frame: Week 65
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Inotersen 300 mg IM Negative | Inotersen 300 mg IM Positive
Number analyzed (Participants) | 4 | 3
L/hr | 3.33 (1.21) | 5.46 (5.13)

ADVERSE EVENTS:
Time Frame: Week 1 to Week 91
Description: Adverse events that first occurred or worsened after the first dose of study drug (inotersen or placebo), including serious adverse events, were summarized for each treatment group. Analysis is based on data collected while study treatment was administered and during follow-up until the day of the participant's last contact date within the study. For each treatment, a participant is counted only once within each preferred term.
Arm/Group | Inotersen | Placebo
All-Cause Mortality (participants affected / at risk) | 5/112 | 0/60
Serious Adverse Events (participants affected / at risk) | 36/112 | 13/60
Other Adverse Events (participants affected / at risk) | 110/112 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotersen (N=112) | Placebo (N=60)
Pneumonia (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 2
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Sinus arrest (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Glomerulonephritis (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Angiopathy (Vascular disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inotersen (N=112) | Placebo (N=60)
Anaemia (Blood and lymphatic system disorders) | 15 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 3
Blepharitis (Eye disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 27 | 12
Dry mouth (Gastrointestinal disorders) | 6 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 15 | 6
Nausea (Gastrointestinal disorders) | 35 | 7
Vomiting (Gastrointestinal disorders) | 17 | 2
Asthenia (General disorders) | 14 | 8
Chills (General disorders) | 20 | 2
Fatigue (General disorders) | 28 | 12
Gait disturbance (General disorders) | 6 | 5
Injection site bruising (General disorders) | 8 | 2
Injection site erythema (General disorders) | 35 | 0
Injection site pain (General disorders) | 23 | 4
Injection site pruritus (General disorders) | 13 | 0
Injection site reaction (General disorders) | 6 | 0
Injection site swelling (General disorders) | 6 | 0
Influenza like illness (General disorders) | 9 | 2
Oedema (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 21 | 6
Pain (General disorders) | 2 | 5
Pyrexia (General disorders) | 22 | 5
Peripheral swelling (General disorders) | 7 | 0
Seasonal allergy (Immune system disorders) | 1 | 4
Urinary tract infection (Infections and infestations) | 21 | 11
Nasopharyngitis (Infections and infestations) | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Influenza (Infections and infestations) | 4 | 3
Rhinitis (Infections and infestations) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 19 | 13
Contusion (Injury, poisoning and procedural complications) | 9 | 1
Thermal burn (Injury, poisoning and procedural complications) | 6 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3
Glomerular filtration rate decreased (Investigations) | 6 | 2
Platelet count decreased (Investigations) | 12 | 0
Weight decreased (Investigations) | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 11 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 8
Headache (Nervous system disorders) | 26 | 7
Paraesthesia (Nervous system disorders) | 11 | 2
Dizziness (Nervous system disorders) | 14 | 7
Syncope (Nervous system disorders) | 9 | 2
Hypoaesthesia (Nervous system disorders) | 10 | 6
Presyncope (Nervous system disorders) | 6 | 0
Neuralgia (Nervous system disorders) | 3 | 8
Neuropathy peripheral (Nervous system disorders) | 2 | 4
Depression (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 6 | 3
Anxiety (Psychiatric disorders) | 1 | 4
Proteinuria (Renal and urinary disorders) | 7 | 2
Haematuria (Renal and urinary disorders) | 5 | 5
Dysuria (Renal and urinary disorders) | 2 | 4
Urinary retention (Renal and urinary disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 | 4
Hypotension (Vascular disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT01737398/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT01737398/SAP_001.pdf